CLINICAL TRIAL: NCT01480427
Title: Assessment of Quality of Life in Food Allergic Children
Status: Completed | Type: Observational
Sponsor: Jacqueline Wassenberg (Other)
Responsible Party: Sponsor-Investigator, Jacqueline Wassenberg, Dr (MD), University of Lausanne Hospitals
Organization: University of Lausanne Hospitals (Other)
Other Study IDs: PedQLFA1
Record Dates: First submitted 2011-11-23; First posted 2011-11-28 (Estimated); Last update posted 2011-11-28 (Estimated); Status verified 2011-11

CONDITIONS: Food Allergy
Keywords: Children aged 0-12 years; IgE mediated food allergy
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
The purpose of this study is

1. To validate in french quality of life questionnaires for food allergic children
2. To evaluate if the quality of life of food allergic french speaking children aged 0-12 years is affected by their condition
3. To validate a didactic game for food allergic children

ELIGIBILITY:
Inclusion Criteria:

* French speaking children with confirmed IgE mediated food allergy
* Aged 0-12 years old

Exclusion Criteria:

* Inclusion in another trial
* Chronic severe diseases

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: General population of children 0-12 years old
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2009-05; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Wassenberg, MD, Principal Investigator — University of Lausanne Hospitals

REFERENCES:
- [Derived] Wassenberg J, Cochard MM, Dunngalvin A, Ballabeni P, Flokstra-de Blok BM, Newman CJ, Hofer M, Eigenmann PA. Parent perceived quality of life is age-dependent in children with food allergy. Pediatr Allergy Immunol. 2012 Aug;23(5):412-9. doi: 10.1111/j.1399-3038.2012.01310.x. Epub 2012 May 3. PMID 22554401